CLINICAL TRIAL: NCT03293459
Title: Influence of Shunt Occlusion on Organ Functions in Hyperammonemic Patients With Cirrhosis Having Porto-systemic Shunt. A Randomized Controlled Trial.
Brief Title: Influence of Shunt Occlusion on Organ Functions in Hyperammonemic Patients With Cirrhosis Having Porto-systemic Shunt.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-13
Record Dates: First submitted 2017-07-03; First posted 2017-09-26 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shunt Occlusion +SMT (Experimental): Shunt Occlusion +SMT
  Interventions: Procedure: Shunt Occlusion; Dietary Supplement: Standard Medical Treatment (SMT)
- Standard Medical Treatment (SMT) (Active Comparator)
  Interventions: Dietary Supplement: Standard Medical Treatment (SMT)

INTERVENTIONS:
Procedure: Shunt Occlusion — Catheterization of the Porto-systemic shunt (via the left renal vein for gastro-lienorenal shunt) will be accomplished using a catheter and occlusion will be performed with balloon catheter/vascular plug. Occlusion venography is then performed to define the type of varix/varices and the anatomy of the venous drainage followed by infusion of sclerosant. The occluded balloon were inflated and remained in place for a maximum of 24 hours deflated under fluoroscopy the next day/plug is deployed and sclerosant is injected to obliterate the shunt and follow up CT is done to look for completion on the next day. Follow up CT abdomen is done periodically to look for effect on shunt and organ.
  Arms: Shunt Occlusion +SMT
Dietary Supplement: Standard Medical Treatment (SMT) — These will include diet rich in BCAA (branch chain amino acids), laxatives and rifaximin

SUMMARY:
The spontaneous Porto-systemic shunt is occluded by intervention procedures like Balloon Occluded Retrograde Transvenous Obliteration (BRTO), Plug-assisted Retrograde Transvenous Obliteration (PARTO) and shunt occlusion procedures resulting in diversion of blood flow towards the portal circulation and in turn the liver. According to this investigator hypothesized that shunt occlusion improves liver volume and function along with beneficial effect on other organ systems by decreasing ammonia and improving hepatopetal flow. All patients with cirrhosis having large shunt(>10mm) and raised ammonia levels and will be randomized to receive standard medical treatment and those receiving shunt occlusion procedures. Investigator will assess organ functions and liver regenerative potential pre and post (after 3 to 15 months) procedure.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the study
* Age 18 to 70 years
* Cirrhotic patients with large shunts (>10mm) and hyperammonemia (arterial ammonia >1.5 x N)

Exclusion Criteria:

* Intractable ascites
* Hepatocellular Carcinoma
* Portal Vein Thrombosis or splenic vein thrombosis
* High risk esophageal varices
* Pregnant and lactation
* Significant heart or respiratory failure
* Active gastrointestinal bleeding
* Refusal to participate in study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Increase in liver volume by CT Volumetry. | 3 to 15 months

SECONDARY OUTCOMES:
Reduction in MELD (Model for End Stage Liver Disease) in both groups | 3 to 15 months
Improvement in T Score | 3 to 15 months
Reduction in Plasma ammonia levels in both groups | 3 to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Amar Mukund, MD, Study Director — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mukund A, Choudhury SP, Tripathy TP, Ananthashayana VH, Jagdish RK, Arora V, Singh SP, Mishra AK, Sarin SK. Influence of shunt occlusion on liver volume and functions in hyperammonemic cirrhosis patients having large porto-systemic shunts: a randomized control trial. Hepatol Int. 2023 Feb;17(1):150-158. doi: 10.1007/s12072-022-10418-4. Epub 2022 Sep 12. PMID 36094625